CLINICAL TRIAL: NCT06469632
Title: Efficacy of Radiofrequency and the Treatment of Myofascial Pain Syndrome in Postpartum Pelvic Pain: Mixed Research Study
Brief Title: Radiofrequency and Myofascial Pain Syndrome in Postpartum Pelvic Pain
Acronym: RASDOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Beatriz Navarro Brazález, Assistant PhD Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/00201/001
Record Dates: First submitted 2023-12-07; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: To be Approved by the Ethics Committee
Keywords: Pelvic Pain; Physiotherapy; Therapeutic adherence; Postpartum; Pelvic floor; Radiofrequency; Myofascial Pain Syndrome
MeSH Terms: conditions — Pelvic Pain; Treatment Adherence and Compliance; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Active Comparator): There will be 12 individual sessions guided by a physiotherapist specialized in Women's Health. The approximate duration will be 45 minutes/session, 2 times a week for 6 weeks. The intervention will consist of a multimodal physiotherapy treatment based on therapeutic patient education, specific PFM exercises, and conservative and invasive treatment of the MPS. Pre- and post-intervention assessments will be carried out, and at 3 and 6 months after the intervention, by an examining physiotherapist who will be blinding for the intervention group.
  Interventions: Other: Active Comparator: Experimental Group 1
- Experimental Group 2 (Experimental): There will be 12 individual sessions guided by a physiotherapist specialized in Women's Health. The approximate duration will be 45 minutes/session, 2 times a week for 6 weeks. The intervention will consist of a multimodal physiotherapy treatment based on therapeutic patient education, specific PFM exercises, conservative and invasive treatment of the MPS and non-ablative radiofrequency. Pre- and post-intervention assessments will be carried out, and at 3 and 6 months after the intervention, by an examining physiotherapist who will be blinding for the intervention group.
  Interventions: Other: Experimental: Experimental Group 2

INTERVENTIONS:
Other: Active Comparator: Experimental Group 1 — Multimodal physiotherapy treatment composed of:
  Therapeutic education about anatomy, physiology and pathophysiology of the abdomino-pelvic cavity, pelvic floor dysfunctions and risk factors, the concept of pain and its associated factors, as well as individual strategies to manage pain.
  Specific PFM exercises performing different types of contractions aimed at improving proprioception, strength, resistance and relaxation capacity.
  Conservative and invasive treatment of MPS active myofascial trigger points (MTP) will be treated by dry needling and Swiss technique. Latent MTP will be treated using the Swiss technique.
  Arms: Experimental Group 1
Other: Experimental: Experimental Group 2 — Multimodal physiotherapy treatment composed of:
  Therapeutic education about anatomy, physiology and pathophysiology of the abdomino-pelvic cavity, pelvic floor dysfunctions and risk factors, the concept of pain and its associated factors, as well as individual strategies to manage pain.
  Specific PFM exercises performing different types of contractions aimed at improving proprioception, strength, resistance and relaxation capacity.
  Conservative and invasive treatment of MPS active myofascial trigger points (MTP) will be treated by dry needling and Swiss technique. Latent MTP will be treated using the Swiss technique.
  Non-ablative radiofrequency: using capacitive superficial electrodes and resistive superficial and intravaginal electrodes.
  Arms: Experimental Group 2

SUMMARY:
About 30% of women experience pain in the perineum and pelvic region one year after the vaginal labor, rising up to 50% when it is triggered during vaginal penetration, called this pain as dyspareunia. An early physiotherapy treatment could be the solution to the pain relief of these women. Thus, the objectives of the present randomised clinical trail are (i) to determine the effectiveness of a physiotherapy treatment based on education therapeutic, the treatment of myofascial pain syndrome (MPS) of the pelvic floor muscles (PFM), and PFM specific training with or without radiofrequency in reducing pain and improving sexual function; and, (ii) to know the facilitating factors and barriers in adherence and perceived self-efficacy towards physiotherapy treatment of women with pelviperineal pain in the postpartum.

Methodology: randomized clinical trial with examinator blinding and two parallel groups, followed by a qualitative study. Thirty eight women per group will be needed with postpartum pelviperineal pain between 8 weeks after labour, with intensity ≥ 4 cm on the visual analogue scale. The assignment will be random to an Experimental 1 group based on therapeutic education, plus conservative and invasive treatment of MPS and specific PFM exercise versus an Experimental 2 group consisted in the same treatment plus non-ablative radiofrequency treatment. In both cases, 12 individual supervised sessions will be held by a physiotherapist specialized in women's health, with evaluations pre- and post-intervention, at 3 and 6 months. The outcome variables will be the intensity of the pain, the presence of MPS at PFM, the PFM contraction quality, sexual function and specific quality of life. The qualitative study will be carried out in the assessment 6 months post-intervention, through interviews semi-structured and focus groups. The interviews will be guided with previous questions established, recorded, transcribed and thematically analyzed by a panel of experts.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women
* Eutocic vaginal birth
* Postpartum pelviperineal pain 8 weeks after birth
* Intensity ≥ 4 cm in the VAS
* Freely signed the Informed consent

Exclusion Criteria:

* Multiparous women
* Instrumental delivery
* Cesarean delivery
* Avulsion of the levator ani muscle
* Diagnosis of coccygodynia and/or coccygeal pain
* Sphincter anal injury during vaginal birth
* History of pelvic fractures and/or neoplasms
* Pregnant women
* Neurological diseases
* Vaginal infection or active urinary tract, or with any
* Uterine device with metallic components
* Women with cognitive, auditory and/or visual limitations to understand information, respond to questionnaires, consent and/or participate in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Pain intensity through the Verbal Numerical Scale (0 no pain, and 10 the most bearable pain) | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  intensity, behavior and location (pain body chart).
Sexual function | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Self-completion of the FSFI questionnaire, which evaluates sexual function based on 6 domains: desire, excitement, lubrication, orgasm, satisfaction and pain. The maximum score is 36, considering sexual dysfunction a value >27.

SECONDARY OUTCOMES:
Pelvic floor dysfunction symptoms | Pre-treatment, post-treatment (after 12 sessions of physiotherapy treatment which will last approximately 3 months after starting the study), 3 and 6 months after treatment
  Presence of urinary, intestinal and/or symptoms suggestive of prolapse
PFM capacity of contraction through Modified Oxford Scale (0 no contraction, 5 strong contraction) | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Intravaginal palpation of pelvic floor muscles with one or two fingers.
PFM capacity of relaxation (yes or no) | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Intravaginal palpation of pelvic floor muscles with one or two fingers.
PFM basal tone in grams | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Intravaginal dynamometry
PFM muscle strength in grams | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Intravaginal dynamometry
Distance of the urogenital hiatus in milimeters | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Assessment through transperineal ultrasound of the distance of the urogenital hiatus at rest, during a strong PFM contraction and during a pushing effort.
Presence of MPS in PFM and abdominal muscles | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Following the diagnostic criteria of Travel and Simons.
Specific quality of life and impact of Pelvoc floor Disfunction using questionnaires: PFDI-20 and PFIQ-7 | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Through the questionnaires: Pelvic Floor Distress Inventory short version (PFDI-20) and Pelvic Floor Impact Questionnaire short form (PFIQ-7). In both questionnaires, the scores range between 0 and 300, where a higher score indicates more distress and more impact on quality of life.
Self-efficacy | Pre-treatment, post-treatment (6 weeks after starting the study), 3 and 6 months after treatment
  Through Broome Pelvic Muscle Self-Efficacy Scale. The score ranges from 0 to 100, where 100 implies greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Navarro-Brazález, PhD, Principal Investigator — Physiotherapy in Women's Health (FPSM) Research Group. Physiotherapy Department, Faculty of Medicine and Health Sciences, University of Alcalá, Alcalá de Henares, 28805 Madrid, Spain.
Locations (1):
- Physiotherapy in Women's Health (FPSM) Research Group. Physiotherapy Department, Faculty of Medicine and Health Sciences, University of Alcalá, Alcalá de Henares, 28805 Madrid, Spain., Alcalá de Henares, Madrid, Spain